CLINICAL TRIAL: NCT02657499
Title: Post Affordable Care Act: Evaluation of Community Health Centers
Brief Title: Post Affordable Care Act Evaluation
Acronym: PACE
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: OCHIN, Inc. (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jennifer E DeVoe, MD DPhil, Principle Investigator, Oregon Health and Science University
Other Study IDs: ARQHR01HS024270
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Chronic Disease
Keywords: healthcare access; utilization; expenditures; preventive services
MeSH Terms: conditions — Chronic Disease; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Medicaid Expansion States: Patients receiving care in community health centers in states that expanded Medicaid (intervention group)
  Interventions: Other: Medicaid Expansion
- Non Medicaid Expansion States: Patients receiving care in community health centers in states that did not expand Medicaid (control group)
  Interventions: Other: Medicaid Expansion

INTERVENTIONS:
Other: Medicaid Expansion — There will be no direct intervention, but rather an observation of change based on whether a state expanded Medicaid or not

SUMMARY:
This innovative study will measure the impact of Affordable Care Act-sponsored Medicaid expansions on access to and utilization of community health center (CHC) services. Building on the investigators prior work that developed a robust community-based research infrastructure within the OCHIN community health information network, the investigator will utilize linked electronic health record data from the OCHIN network of >400 CHC clinics in 8 states that expanded Medicaid coverage and 8 states that did not expand.

DETAILED DESCRIPTION:
The Affordable Care Act (ACA) called for every state in the United States (US) to expand Medicaid coverage to individuals at ≤138% of the federal poverty level by 2014. In a 2012 legal challenge, the Supreme Court ruled that states were not required to implement the ACA-sponsored Medicaid expansion; thus (by December 31, 2014), only 27 states and the District of Columbia expanded Medicaid, while 23 states did not. Little is known about the impact of ACA-sponsored Medicaid expansions on access to and changes in receipt of healthcare services among vulnerable populations. Yet this knowledge is essential to informing deliberations in 'non-expansion' states regarding whether to expand their Medicaid programs, and will also be helpful to 'expansion' states eager to learn about the impact of their expansions. The natural experiment created by the Supreme Court decision to make expansion optional for states provides a unique opportunity to assess the extent to which Medicaid expansions improve access to healthcare for low-income patients and other vulnerable populations. The proposed project will be one of the first to examine changes in access to and receipt of healthcare services and to Medicaid expenditures following ACA Medicaid expansions among a large population of safety net clinic patients. The investigators will use electronic health record data (EHR) from the OCHIN practice-based research network, which serves >1 million patients in 442 community health centers (CHCs) in 8 expansion states and 8 non-expansion states. Moreover, using CHC data from the 8 expansion-states, the investigators will examine differences in utilization among patients gaining new Medicaid coverage (newly insured), as compared to those already insured by Medicaid (already insured), and those who remain uninsured (uninsured). Finally, the investigators will link EHR data from the 213 OCHIN clinics in Oregon to Medicaid administrative claims data to assess overall healthcare utilization (including care received outside of CHCs, such as hospitalization) and to compare Medicaid expenditures among newly insured individuals versus those already insured. The investigators will address the following specific aims: Aim 1: compare pre-post health insurance status, primary care, mental health, and dental visits, and receipt of preventive services, as well as changes in payer mix among OCHIN CHCs in states that did and did not expand Medicaid; Aim 2: Examine pre-post utilization of CHC services (including receipt of preventive services) by newly insured patients compared to already insured patients and uninsured patients; and, Aim 3: Measure pre-post Medicaid expansion changes in overall utilization of healthcare services and costs to the Oregon Medicaid program among newly insured compared to already insured. The findings from this project will be extremely relevant to policy and practice, informing further improvements in the US healthcare system to ensure access to healthcare for vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients in intervention and control states aged 20-64

Exclusion Criteria:

* Patients outside of age range 20-64

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study eligible patients within electronic health record data from the OCHIN community health information network
Sampling Method: Non-Probability Sample
Enrollment: 1939848 (Actual)
Dates: Start 2012-01; Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Health Insurance Status | 24 months prior to Medicaid expansion vs 24 months post
  Health insurance status derived from EHR data and is primarily based on information collected at each visit

SECONDARY OUTCOMES:
Healthcare service utilization | 24 months prior to Medicaid expansion vs 24 months post
  Number and type of internal services utilized
Preventive Service utilization | 24 months prior to Medicaid expansion vs 24 months post
  Number and type of preventive services received
Medicaid Expenditures | 24 months prior to Medicaid expansion vs 24 months post
  We will calculate the average pre-post expansion difference in total Medicaid expenditures. We will attach an expenditure for each service based on its average Medicaid Fee-For-Service reimbursement in the first year for those who were insured or uninsured pre or post expansion

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E DeVoe, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marino M, Angier H, Valenzuela S, Hoopes M, Killerby M, Blackburn B, Huguet N, Heintzman J, Hatch B, O'Malley JP, DeVoe JE. Medicaid coverage accuracy in electronic health records. Prev Med Rep. 2018 Jul 27;11:297-304. doi: 10.1016/j.pmedr.2018.07.009. eCollection 2018 Sep. PMID 30116701
- [Result] Hoopes MJ, Angier H, Gold R, Bailey SR, Huguet N, Marino M, DeVoe JE. Utilization of Community Health Centers in Medicaid Expansion and Nonexpansion States, 2013-2014. J Ambul Care Manage. 2016 Oct-Dec;39(4):290-8. doi: 10.1097/JAC.0000000000000123. PMID 26765808
- [Result] Springer R, Marino M, O'Malley JP, Lindner S, Huguet N, DeVoe JE. Oregon Medicaid Expenditures After the 2014 Affordable Care Act Medicaid Expansion: Over-time Differences Among New, Returning, and Continuously Insured Enrollees. Med Care. 2018 May;56(5):394-402. doi: 10.1097/MLR.0000000000000907. PMID 29578955
- [Result] Angier, H., C. J. Tillotson, L. S. Wallace, M. Marino, J. P. O' Malley, A. Sumic, L. Baker, C. Nelson, N. Huguet, A. Suchocki, H. Holderness and J. E. DeVoe (2018).
- [Result] Angier H, Hoopes M, Marino M, Huguet N, Jacobs EA, Heintzman J, Holderness H, Hood CM, DeVoe JE. Uninsured Primary Care Visit Disparities Under the Affordable Care Act. Ann Fam Med. 2017 Sep;15(5):434-442. doi: 10.1370/afm.2125. PMID 28893813
- [Result] Huguet N, Hoopes MJ, Angier H, Marino M, Holderness H, DeVoe JE. Medicaid Expansion Produces Long-Term Impact on Insurance Coverage Rates in Community Health Centers. J Prim Care Community Health. 2017 Oct;8(4):206-212. doi: 10.1177/2150131917709403. Epub 2017 May 17. PMID 28513249
- [Result] Heintzman J, Bailey SR, DeVoe J, Cowburn S, Kapka T, Duong TV, Marino M. In Low-Income Latino Patients, Post-Affordable Care Act Insurance Disparities May Be Reduced Even More than Broader National Estimates: Evidence from Oregon. J Racial Ethn Health Disparities. 2017 Jun;4(3):329-336. doi: 10.1007/s40615-016-0232-1. Epub 2016 Apr 22. PMID 27105630
- [Result] Hatch B, Marino M, Killerby M, Angier H, Hoopes M, Bailey SR, Heintzman J, O'Malley JP, DeVoe JE. Medicaid's Impact on Chronic Disease Biomarkers: A Cohort Study of Community Health Center Patients. J Gen Intern Med. 2017 Aug;32(8):940-947. doi: 10.1007/s11606-017-4051-9. Epub 2017 Apr 3. PMID 28374214
- [Result] Bailey SR, Hoopes MJ, Marino M, Heintzman J, O'Malley JP, Hatch B, Angier H, Fortmann SP, DeVoe JE. Effect of Gaining Insurance Coverage on Smoking Cessation in Community Health Centers: A Cohort Study. J Gen Intern Med. 2016 Oct;31(10):1198-205. doi: 10.1007/s11606-016-3781-4. Epub 2016 Jun 21. PMID 27329121

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Statistical Analysis Plan only (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT02657499/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan only (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT02657499/SAP_001.pdf